CLINICAL TRIAL: NCT00452764
Title: Phenotype and Number of Regulatory T Cells Present in Peripheral Blood of COPD Patients Versus Healthy Controls
Brief Title: Regulatory T Cells in COPD
Status: Completed | Type: Observational
Sponsor: Groningen Research Institute for Asthma and COPD (Other)
Other Study IDs: METc2006-135
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Healthy; Regulatory T cell; Heme oxygenase-1; peripheral blood
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Withdrawal of medication

SUMMARY:
Lymphoid follicles, consisting of T-and B cells, are involved in the chronic inflammatory response in COPD. Foxp3 positive regulatory T cells (Tregs) are present in these follicles and may be involved in the suppression of this chronic inflammatory response.

We hypothesise that a dysfunction of Tregs underlies the development of the inflammatory response in COPD. This could be either due to a decreased presence of Tregs in COPD, or to an altered function of Tregs possibly caused by a decreased HO-1 expression and/or an altered TGFβ regulation.

DETAILED DESCRIPTION:
COPD is a leading cause of death worldwide and its morbidity and mortality are still rising.So far, no effective treatment is available To find better treatment methods more insight is needed in the nature/origin of the chronic inflammation that underlies the development of COPD.

The important role of neutrophils, macrophages and cytotoxic T cells is well established in this respect, yet the role of CD4 T cells and B cells has only recently (re)attracted attention. We detected the presence of lymphoid follicles in lung tissue of COPD patients, consisting of B cells surrounded by T cells. Recently, we have found the presence of Foxp3 positive T cells as a component of these lymphoid follicles in COPD. Since Foxp3 is a distinctive marker of regulatory T cells (Tregs), this finding suggests that Tregs are involved in the inflammatory response in COPD.

Tregs are important in controlling immunological tolerance and preventing auto-immune responses by inhibiting T-cell responses. Dysfunction of Tregs can lead to auto-immune diseases, allergy and chronic inflammatory diseases. However, nothing is known so far about their contribution to the chronic inflammatory response in COPD. Recent studies show that, next to direct inhibition by cell-cell contact, the inhibitory effects of Tregs are mediated by heme oxygenase-1 (HO-1) expression and membrane bound TGFβ.

We hypothesise that a dysfunction of regulatory T cells underlies the development of the inflammatory response in COPD. This could be due to a decreased presence of Tregs in COPD, or to an altered function of Tregs. The latter may be due to a decreased HO-1 expression, as we have shown in macrophages of COPD patients compared to those in healthy controls, and/or an altered TGFβ regulation, a cytokine that plays a prime role in COPD.

ELIGIBILITY:
Inclusion Criteria:

COPD patients

* Clinical diagnosed COPD
* No allergies
* Post-bronchodilator FEV1 < 80% predicted, and post-bronchodilator FEV1/FVC < 70%
* No use of (inhaled) corticosteroids in the 6 weeks preceding the study
* Age > 40
* Smokers and ex- smokers > 10 pack years
* Ex-smokers have to have quitted smoking for at least one year
* No other major current health problems
* Informed consent Healthy controls
* No signs of pulmonary disease
* No allergies or hyperreactivity
* No other major current health problems
* FEV1 > 90 % predicted, FEV1/FVC > 70%
* Age > 40
* Never smokers, i.e. no cigarettes last year, and maximal 5 pack years
* Smokers and ex- smokers > 10 pack years
* Ex-smokers have to have quitted smoking for at least one year
* Informed consent

Exclusion Criteria:

* Use of (inhaled) corticosteroids in the 6 weeks preceding the study
* Addiction to alcohol or drugs
* COPD exacerbation in the 6 weeks preceding the study

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huib AM Kerstjens, MD, PhD, Principal Investigator — UMCG, department of pulmonary diseases
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands